CLINICAL TRIAL: NCT04513054
Title: Is There a Genetic Predisposition for Acute Stress-induced (Takotsubo) Cardiomyopathy: The GENETIC Study
Brief Title: Is There a Genetic Predisposition for Acute Stress-induced (Takotsubo) Cardiomyopathy
Acronym: GENETIC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aberdeen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2-025-18
Record Dates: First submitted 2020-08-03; First posted 2020-08-14 (Actual); Last update posted 2024-12-24 (Actual); Status verified 2024-12

CONDITIONS: Takotsubo Cardiomyopathy
MeSH Terms: conditions — Takotsubo Cardiomyopathy | interventions — Genetic Testing

STUDY DESIGN:
Intervention Model Description: Single group observational study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Takotsubo Case Arm (Other): A patient that has been diagnosed with Takotsubo Cardiomyopathy from 2010 onwards.
  Interventions: Genetic: Blood collection for genetic analysis

INTERVENTIONS:
Genetic: Blood collection for genetic analysis — Blood collection for genetic analysis

SUMMARY:
Acute stress-induced (takotsubo) cardiomyopathy or broken heart syndrome presents like a heart attack, classically is triggered by intense emotional or physical stress and can have serious health consequences. In the current study the investigators wish to establish whether there is a genetic predisposition making certain people more susceptible to this condition. This could also have implications for their families.

DETAILED DESCRIPTION:
Acute stress-induced (takotsubo) cardiomyopathy presents like a myocardial infarct, is triggered by intense emotional or physical stress, and can have catastrophic and potentially fatal consequences. Despite data linking takotsubo cardiomyopathy with conditions that have a recognized genetic predisposition (such as mental health and neurological problems), a systematic and comprehensive characterisation of the genetic-epidemiologic factors in takotsubo is lacking. The researchers propose to further investigate this disorder by collecting blood from probands and characterising the genotype of patients with takotsubo cardiomyopathy in a large scale, nationwide genome wide association study. The investigators will also archive DNA for identification of future candidate genetic variants. Ultimately, understanding the underlying predisposition of this poorly understood neuro-psycho-cardiac disorder is essential if we are to move this field forward.

ELIGIBILITY:
Inclusion Criteria:

* All patients who have been diagnosed with Takotsubo cardiomyopathy in Scotland between 2010 to date.
* Familial cases elsewhere in the world who would be willing to participate.

Exclusion Criteria:

* Unwillingness to participate

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 700 (Estimated)
Dates: Start 2019-03-12 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Genome Wide Association Study | At baseline
  Genome Wide Association Study to search for susceptibility variants

CONTACTS AND LOCATIONS:
Overall Officials: Dana K Dawson, MD, MPhil, Principal Investigator — University of Aberdeen
Locations (1):
- Cardiovascular Research Facility, Aberdeen, Aberdeenshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Prasad A, Lerman A, Rihal CS. Apical ballooning syndrome (Tako-Tsubo or stress cardiomyopathy): a mimic of acute myocardial infarction. Am Heart J. 2008 Mar;155(3):408-17. doi: 10.1016/j.ahj.2007.11.008. Epub 2008 Jan 31. PMID 18294473
- [Background] Templin C, Ghadri JR, Diekmann J, Napp LC, Bataiosu DR, Jaguszewski M, Cammann VL, Sarcon A, Geyer V, Neumann CA, Seifert B, Hellermann J, Schwyzer M, Eisenhardt K, Jenewein J, Franke J, Katus HA, Burgdorf C, Schunkert H, Moeller C, Thiele H, Bauersachs J, Tschope C, Schultheiss HP, Laney CA, Rajan L, Michels G, Pfister R, Ukena C, Bohm M, Erbel R, Cuneo A, Kuck KH, Jacobshagen C, Hasenfuss G, Karakas M, Koenig W, Rottbauer W, Said SM, Braun-Dullaeus RC, Cuculi F, Banning A, Fischer TA, Vasankari T, Airaksinen KE, Fijalkowski M, Rynkiewicz A, Pawlak M, Opolski G, Dworakowski R, MacCarthy P, Kaiser C, Osswald S, Galiuto L, Crea F, Dichtl W, Franz WM, Empen K, Felix SB, Delmas C, Lairez O, Erne P, Bax JJ, Ford I, Ruschitzka F, Prasad A, Luscher TF. Clinical Features and Outcomes of Takotsubo (Stress) Cardiomyopathy. N Engl J Med. 2015 Sep 3;373(10):929-38. doi: 10.1056/NEJMoa1406761. PMID 26332547
- [Background] Stiermaier T, Moeller C, Oehler K, Desch S, Graf T, Eitel C, Vonthein R, Schuler G, Thiele H, Eitel I. Long-term excess mortality in takotsubo cardiomyopathy: predictors, causes and clinical consequences. Eur J Heart Fail. 2016 Jun;18(6):650-6. doi: 10.1002/ejhf.494. Epub 2016 Mar 14. PMID 26990821
- [Background] Sy F, Basraon J, Zheng H, Singh M, Richina J, Ambrose JA. Frequency of Takotsubo cardiomyopathy in postmenopausal women presenting with an acute coronary syndrome. Am J Cardiol. 2013 Aug 15;112(4):479-82. doi: 10.1016/j.amjcard.2013.04.010. Epub 2013 May 16. PMID 23683950
- [Background] Scally C, Ahearn T, Rudd A, Neil CJ, Srivanasan J, Jagpal B, Horowitz J, Frenneaux M, Dawson DK. Right Ventricular Involvement and Recovery After Acute Stress-Induced (Tako-tsubo) Cardiomyopathy. Am J Cardiol. 2016 Mar 1;117(5):775-80. doi: 10.1016/j.amjcard.2015.11.057. Epub 2015 Dec 13. PMID 26782339
- [Background] Dawson DK, Neil CJ, Henning A, Cameron D, Jagpal B, Bruce M, Horowitz J, Frenneaux MP. Tako-Tsubo Cardiomyopathy: A Heart Stressed Out of Energy? JACC Cardiovasc Imaging. 2015 Aug;8(8):985-7. doi: 10.1016/j.jcmg.2014.10.004. Epub 2014 Nov 1. No abstract available. PMID 25499134
- [Background] Scally C, Rudd A, Mezincescu A, Wilson H, Srivanasan J, Horgan G, Broadhurst P, Newby DE, Henning A, Dawson DK. Persistent Long-Term Structural, Functional, and Metabolic Changes After Stress-Induced (Takotsubo) Cardiomyopathy. Circulation. 2018 Mar 6;137(10):1039-1048. doi: 10.1161/CIRCULATIONAHA.117.031841. Epub 2017 Nov 11. PMID 29128863
- [Background] Tornvall P, Collste O, Ehrenborg E, Jarnbert-Petterson H. A Case-Control Study of Risk Markers and Mortality in Takotsubo Stress Cardiomyopathy. J Am Coll Cardiol. 2016 Apr 26;67(16):1931-6. doi: 10.1016/j.jacc.2016.02.029. PMID 27102508
- [Background] Sharkey SW, Maron BJ. Epidemiology and clinical profile of Takotsubo cardiomyopathy. Circ J. 2014;78(9):2119-28. doi: 10.1253/circj.cj-14-0770. Epub 2014 Aug 5. PMID 25099475
- [Background] Pison L, De Vusser P, Mullens W. Apical ballooning in relatives. Heart. 2004 Dec;90(12):e67. doi: 10.1136/hrt.2004.046813. PMID 15547001
- [Background] Kumar G, Holmes DR Jr, Prasad A. "Familial" apical ballooning syndrome (Takotsubo cardiomyopathy). Int J Cardiol. 2010 Oct 29;144(3):444-5. doi: 10.1016/j.ijcard.2009.03.078. Epub 2009 Apr 17. PMID 19375184
- [Background] Sharkey SW, Lips DL, Pink VR, Maron BJ. Daughter-mother tako-tsubo cardiomyopathy. Am J Cardiol. 2013 Jul 1;112(1):137-8. doi: 10.1016/j.amjcard.2013.02.063. Epub 2013 Apr 2. PMID 23561588
- [Background] Caretta G, Robba D, Vizzardi E, Bonadei I, Raddino R, Metra M. Tako-tsubo cardiomyopathy in two sisters: a chance finding or familial predisposition? Clin Res Cardiol. 2015 Jul;104(7):614-6. doi: 10.1007/s00392-015-0837-0. Epub 2015 Mar 6. No abstract available. PMID 25743177
- [Background] Ikutomi M, Yamasaki M, Matsusita M, Watari Y, Arashi H, Endo G, Yamaguchi J, Ohnishi S. Takotsubo cardiomyopathy in siblings. Heart Vessels. 2014 Jan;29(1):119-22. doi: 10.1007/s00380-013-0345-y. Epub 2013 Apr 7. PMID 23563753
- [Background] Wittstein IS, Thiemann DR, Lima JA, Baughman KL, Schulman SP, Gerstenblith G, Wu KC, Rade JJ, Bivalacqua TJ, Champion HC. Neurohumoral features of myocardial stunning due to sudden emotional stress. N Engl J Med. 2005 Feb 10;352(6):539-48. doi: 10.1056/NEJMoa043046. PMID 15703419
- [Background] Goodloe AH, Evans JM, Middha S, Prasad A, Olson TM. Characterizing genetic variation of adrenergic signalling pathways in Takotsubo (stress) cardiomyopathy exomes. Eur J Heart Fail. 2014 Sep;16(9):942-9. doi: 10.1002/ejhf.145. Epub 2014 Aug 8. PMID 25132214
- [Background] Figtree GA, Bagnall RD, Abdulla I, Buchholz S, Galougahi KK, Yan W, Tan T, Neil C, Horowitz JD, Semsarian C, Ward MR. No association of G-protein-coupled receptor kinase 5 or beta-adrenergic receptor polymorphisms with Takotsubo cardiomyopathy in a large Australian cohort. Eur J Heart Fail. 2013 Jul;15(7):730-3. doi: 10.1093/eurjhf/hft040. PMID 23794609
- [Background] Sharkey SW, Maron BJ, Nelson P, Parpart M, Maron MS, Bristow MR. Adrenergic receptor polymorphisms in patients with stress (tako-tsubo) cardiomyopathy. J Cardiol. 2009 Feb;53(1):53-7. doi: 10.1016/j.jjcc.2008.08.006. Epub 2008 Oct 9. PMID 19167638
- [Background] Eitel I, Moeller C, Munz M, Stiermaier T, Meitinger T, Thiele H, Erdmann J. Genome-wide association study in takotsubo syndrome - Preliminary results and future directions. Int J Cardiol. 2017 Jun 1;236:335-339. doi: 10.1016/j.ijcard.2017.01.093. Epub 2017 Jan 15. PMID 28108127
- [Background] Nelson CP, Goel A, Butterworth AS, Kanoni S, Webb TR, Marouli E, Zeng L, Ntalla I, Lai FY, Hopewell JC, Giannakopoulou O, Jiang T, Hamby SE, Di Angelantonio E, Assimes TL, Bottinger EP, Chambers JC, Clarke R, Palmer CNA, Cubbon RM, Ellinor P, Ermel R, Evangelou E, Franks PW, Grace C, Gu D, Hingorani AD, Howson JMM, Ingelsson E, Kastrati A, Kessler T, Kyriakou T, Lehtimaki T, Lu X, Lu Y, Marz W, McPherson R, Metspalu A, Pujades-Rodriguez M, Ruusalepp A, Schadt EE, Schmidt AF, Sweeting MJ, Zalloua PA, AlGhalayini K, Keavney BD, Kooner JS, Loos RJF, Patel RS, Rutter MK, Tomaszewski M, Tzoulaki I, Zeggini E, Erdmann J, Dedoussis G, Bjorkegren JLM; EPIC-CVD Consortium; CARDIoGRAMplusC4D; UK Biobank CardioMetabolic Consortium CHD working group; Schunkert H, Farrall M, Danesh J, Samani NJ, Watkins H, Deloukas P. Association analyses based on false discovery rate implicate new loci for coronary artery disease. Nat Genet. 2017 Sep;49(9):1385-1391. doi: 10.1038/ng.3913. Epub 2017 Jul 17. PMID 28714975
- [Background] Nikpay M, Goel A, Won HH, Hall LM, Willenborg C, Kanoni S, Saleheen D, Kyriakou T, Nelson CP, Hopewell JC, Webb TR, Zeng L, Dehghan A, Alver M, Armasu SM, Auro K, Bjonnes A, Chasman DI, Chen S, Ford I, Franceschini N, Gieger C, Grace C, Gustafsson S, Huang J, Hwang SJ, Kim YK, Kleber ME, Lau KW, Lu X, Lu Y, Lyytikainen LP, Mihailov E, Morrison AC, Pervjakova N, Qu L, Rose LM, Salfati E, Saxena R, Scholz M, Smith AV, Tikkanen E, Uitterlinden A, Yang X, Zhang W, Zhao W, de Andrade M, de Vries PS, van Zuydam NR, Anand SS, Bertram L, Beutner F, Dedoussis G, Frossard P, Gauguier D, Goodall AH, Gottesman O, Haber M, Han BG, Huang J, Jalilzadeh S, Kessler T, Konig IR, Lannfelt L, Lieb W, Lind L, Lindgren CM, Lokki ML, Magnusson PK, Mallick NH, Mehra N, Meitinger T, Memon FU, Morris AP, Nieminen MS, Pedersen NL, Peters A, Rallidis LS, Rasheed A, Samuel M, Shah SH, Sinisalo J, Stirrups KE, Trompet S, Wang L, Zaman KS, Ardissino D, Boerwinkle E, Borecki IB, Bottinger EP, Buring JE, Chambers JC, Collins R, Cupples LA, Danesh J, Demuth I, Elosua R, Epstein SE, Esko T, Feitosa MF, Franco OH, Franzosi MG, Granger CB, Gu D, Gudnason V, Hall AS, Hamsten A, Harris TB, Hazen SL, Hengstenberg C, Hofman A, Ingelsson E, Iribarren C, Jukema JW, Karhunen PJ, Kim BJ, Kooner JS, Kullo IJ, Lehtimaki T, Loos RJF, Melander O, Metspalu A, Marz W, Palmer CN, Perola M, Quertermous T, Rader DJ, Ridker PM, Ripatti S, Roberts R, Salomaa V, Sanghera DK, Schwartz SM, Seedorf U, Stewart AF, Stott DJ, Thiery J, Zalloua PA, O'Donnell CJ, Reilly MP, Assimes TL, Thompson JR, Erdmann J, Clarke R, Watkins H, Kathiresan S, McPherson R, Deloukas P, Schunkert H, Samani NJ, Farrall M. A comprehensive 1,000 Genomes-based genome-wide association meta-analysis of coronary artery disease. Nat Genet. 2015 Oct;47(10):1121-1130. doi: 10.1038/ng.3396. Epub 2015 Sep 7. PMID 26343387